CLINICAL TRIAL: NCT05356416
Title: Comparative Effects of Dry Needling and Ischemic Compression Technique on Pain, Disability and Range of Motion With Scalene Myofascial Pain Syndrome
Brief Title: Comparative Effects of Dry Needling and Ischemic Compression Technique on Scalene Myofascial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/22/0113 Arooj
Record Dates: First submitted 2022-04-28; First posted 2022-05-02 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Scalenus Syndrome
Keywords: dry needing; myofascial pain; pain; disability
MeSH Terms: conditions — Pain | interventions — Acupressure; Dry Needling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ischemic compression (Experimental): Patients in Group B will receive a single session of ischemic compression technique for ischemic compression technique sustained pressure on the trigger points will be maintained for 30 seconds.
  Interventions: Other: Ischemic compression
- Dry Needling (Active Comparator): Patients in dry needling (DN) group will receive a single session of DN of 10 minutes with sterile needles insert on trigger points in scalene muscles as first twitch response will obtained needles will be manipulated in and out of the muscles to get 2 or 3 more local responses.
  Interventions: Other: Dry needling

INTERVENTIONS:
Other: Ischemic compression — Ischemic compression technique is a massage technique that consists of moderate compression, typically applied with the fingers, to the MTrP. Application of this technique to an MTrP results in a positive effect on pain-pressure threshold.
  Patients in Group B will receive a single session of ischemic compression technique for ischemic compression technique sustained pressure on the trigger points will be maintained for 30 seconds.
  Arms: Ischemic compression
Other: Dry needling — Trigger-point dry needling is an invasive procedure where a fine needle or acupuncture needle is inserted into the skin and muscle.
  Patients in dry needling (DN) group will receive a single session of DN of 10 minutes with sterile needles insert on trigger points in scalene muscles as first twitch response will obtained needles will be manipulated in and out of the muscles to get 2 or 3 more local responses.
  Arms: Dry Needling

SUMMARY:
Myofascial Pain Syndrome (MPS) is a medical term used to describe chronic regional pain syndrome that presents with hyperirritable spots called trigger points (TPs) and/or tender spots (TSs) that arise from taut bands (TB) in the skeletal muscle. Scalene myofascial pain syndrome is a regional pain syndrome wherein pain originates over the neck area and radiates down to the arm. Functionally, MPS causes the muscle to become weak and stiff, leading to reductions in range of movement. Thus, MPS is known as a major cause of morbidity, with a significant impact on daily activity, function and quality of life. The aim of this study is to compare the effects of dry needling versus ischemic compression technique on trigger points of scalene in neck pain, related disability and neck active range of motion among patients with scalene myofascial pain syndrome.

DETAILED DESCRIPTION:
A Randomized clinical trial will be conducted at DHQ Gujranwala and Sikandar medical complex Gujranwala through convenience sampling technique on 24 patients. Patients with scalene myofascial pain syndrome between age from 18 years to 45 with positive Scalene Cramp Test will be included in study. Patients will be accessed for neck pain, disability and active range of motion. They will be allocated through simple random sampling through sealed opaque envelopes into group A and group B. Patients in dry needling (DN) group will receive a single session of DN with sterile needles insert on trigger points in scalene muscles as first twitch response will obtained needles will be manipulated in and out of the muscles to get 2 or 3 more local responses. Patients in Group B will receive a single session of ischemic compression technique for this ischemic compression technique sustained pressure on the trigger points will be maintained for 30 seconds. Control treatment will be same for both groups. Pre and post treatment values will be identified after one month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with scalene myofascial pain syndrome
* Age from 18 years to 45
* Patients with positive Scalene Cramp Test

Exclusion Criteria:

* Whiplash injury
* Thoracic dysfunction any cervical radiculopathy
* Age below 18 and more than 45 years
* Any psychiatry disorder or
* Any contraindication to Dry Needling

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2022-10-18 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | follow up at 4th week
  The Numeric Pain Rating Scale (NPRS) an outcome measure that is a unidimensional measure of pain intensity in adults, including those with chronic pain.
  The NPRS is a segmented numeric version in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of pain.
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
  The NPRS takes <1 minute to complete The NPRS is a valid and reliable scale to measure pain intensity;
  * High test-retest reliability has been (r = 0.96 and 0.95, respectively)
  * For construct validity, the NPRS was shown to be highly correlated: correlations range from 0.86 to 0.95.
Neck Disability Index (NDI) | follow up at 4th week
  This questionnaire has been designed to give us information as to how your neck pain has affected your ability to manage in everyday life. Every section is marked in each section only the one box that applies to you. We realise you may consider that two or more statements in any one section relate to you, but please just mark the box that most closely describes your problem. Intended population includes: Chronic neck or upper back pain and musculoskeletal neck pain.
  Scoring: For each section the total possible score is 5: if the first statement is marked the section score = 0, if the last statement is marked it = 5. If all ten sections are completed the score is calculated.
Universal Goniometer (UG) | follow up at 4th week
  A goniometer is an instrument that measures the available range of motion at a joint. To measure the range of motion physical therapists most commonly use a goniometer. It is necessary that a single notation system is used in goniometry. The neutral zero method (0 to 180- degree system) is the most widely used method. The same goniometer should always be used to reduce the chances of instrumental error.

CONTACTS AND LOCATIONS:
Overall Officials: samrood Akram, MPhil, Principal Investigator — Riphah International University,Lahore
Locations (1):
- Sikandar Medical Complex, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gohil D, Vaishy S, Baxi G, Samson A, Palekar T. Effectiveness of strain-counterstrain technique versus digital ischemic compression on myofascial trigger points. Archives of Medicine and Health Sciences. 2020;8(2):191.
- [Background] Kisilewicz A, Janusiak M, Szafraniec R, Smoter M, Ciszek B, Madeleine P, Fernandez-de-Las-Penas C, Kawczynski A. Changes in Muscle Stiffness of the Trapezius Muscle After Application of Ischemic Compression into Myofascial Trigger Points in Professional Basketball Players. J Hum Kinet. 2018 Oct 15;64:35-45. doi: 10.2478/hukin-2018-0043. eCollection 2018 Sep. PMID 30429897
- [Background] Ortega-Santiago R, Maestre-Lerga M, Fernandez-de-Las-Penas C, Cleland JA, Plaza-Manzano G. Widespread Pressure Pain Sensitivity and Referred Pain from Trigger Points in Patients with Upper Thoracic Spine Pain. Pain Med. 2019 Jul 1;20(7):1379-1386. doi: 10.1093/pm/pnz020. PMID 30821833
- [Background] Bagcier F, Yurdakul O, Ozduran E. Three Simple Rules in Pectoral Muscle's Trigger Point Treatment, Which May Be a Cause of Chest Pain: Position, Palpation, and Perpendicular Needling. J Am Board Fam Med. 2020 Nov-Dec;33(6):1031. doi: 10.3122/jabfm.2020.06.200342. No abstract available. PMID 33219086
- [Background] Boyce D, Wempe H, Campbell C, Fuehne S, Zylstra E, Smith G, Wingard C, Jones R. ADVERSE EVENTS ASSOCIATED WITH THERAPEUTIC DRY NEEDLING. Int J Sports Phys Ther. 2020 Feb;15(1):103-113. PMID 32089962
- [Background] Nasb M, Qun X, Ruckmal Withanage C, Lingfeng X, Hong C. Dry Cupping, Ischemic Compression, or Their Combination for the Treatment of Trigger Points: A Pilot Randomized Trial. J Altern Complement Med. 2020 Jan;26(1):44-50. doi: 10.1089/acm.2019.0231. Epub 2019 Oct 3. PMID 31580695
- [Background] Maayah MF, Khabour OF, Gaowgzeh RA, Neamatallah Z, Alfawaz SS. Effects of acupressure versus physical therapy on Enkephalin and Endorphin levels in Scalene Myofascial Pain Syndrome patients: A randomized controlled trial. Advances in Mechanics. 2021;9(3):1141-53.
- [Background] Yasar MF, Yaksi E, Kurul R, Alisik T, Seker Z. Comparison of dry needling and kinesio taping methods in the treatment of myofascial pain syndrome: A single blinded randomised controlled study. Int J Clin Pract. 2021 Oct;75(10):e14561. doi: 10.1111/ijcp.14561. Epub 2021 Jul 12. PMID 34159691
- [Background] Toghtamesh M, Tajali SB, Jalaei S. Comparing Between the Effects of Dry Needling and Shock Wave in the Treatment of Trapezius Myofascial Pain. Journal of Modern Rehabilitation. 2020;14(4):225-32.
- [Background] Lamba D. Comparison of two different photobiostimulation on pain and functional ability in patients with myofascial trigger points (levator scapulae muscle). International Journal of Medical Research & Health Sciences. 2019;8(7):22-9.